CLINICAL TRIAL: NCT03347370
Title: Subcutaneous (SC) Interferon Beta Therapy in Multiple Sclerosis Patients and Characterization of Injection Site Reactions and Flu-Like Symptoms Under Daily Practice Setting
Brief Title: A Post-Authorization Safety Study of Interferon Beta Therapy in Participants With Multiple Sclerosis
Acronym: PERFECT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: AMS Advanced Medical Services GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: GER-PEG-16-10988
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: subcutaneous interferon beta therapy multiple sclerosis (MS); injection site reactions (ISR); flu-like symptoms (FLS); non-interventional study (NIS); SC Peginterferon beta-1a; SC interferon beta-1a; SC interferon beta-1b; Plegridy®; Betaferon®; Extavia®; Rebif®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Injection Site Reaction | interventions — peginterferon beta-1a; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SC Peginterferon beta-1a: Participants with relapsing-remitting multiple sclerosis (RRMS), currently stable on SC interferon beta treatment for three months or longer (switch between SC interferon beta treatments possible).
  Interventions: Drug: SC Peginterferon beta-1a
- SC interferon beta-1a: Participants with relapsing-remitting multiple sclerosis (RRMS), currently stable on SC interferon beta treatment for three months or longer (switch between SC interferon beta treatments possible).
  Interventions: Drug: SC interferon beta-1a
- SC interferon beta-1b: Participants with relapsing-remitting multiple sclerosis (RRMS), currently stable on SC interferon beta treatment for three months or longer (switch between SC interferon beta treatments possible).
  Interventions: Drug: SC interferon beta-1b

INTERVENTIONS:
Drug: SC Peginterferon beta-1a — All participants will be treated with their current SC interferon beta medication according to the Fachinformation (German equivalent to summary of product characteristics [SmPC]).
  Other Names: Plegridy
  Groups: SC Peginterferon beta-1a
Drug: SC interferon beta-1a — All participants will be treated with their current SC interferon beta medication according to the Fachinformation (German equivalent to summary of product characteristics [SmPC]).
  Other Names: Rebif
  Groups: SC interferon beta-1a
Drug: SC interferon beta-1b — All participants will be treated with their current SC interferon beta medication according to the Fachinformation (German equivalent to summary of product.
  Other Names: Betaferon; Extavia
  Groups: SC interferon beta-1b

SUMMARY:
The purpose of this study is to investigate the safety of subcutaneous (SC) interferon beta therapies with regard to frequency of injection site reactions (ISR) and flu-like symptoms (FLS) as reported by the relapsing-remitting multiple sclerosis (RRMS) participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose of the study and provide signed and dated informed consent
* Diagnosed relapsing-remitting multiple sclerosis
* Currently receiving a SC interferon beta treatment (label conform)
* Stable on SC interferon beta treatment for three months or longer (switch between SC interferon beta treatments possible).

Key Exclusion Criteria:

* Contraindications according to the Fachinformation (German equivalent to Summary of Product Characteristics [SmPC])
* Treatment with Glatiramer acetate and intramuscular (IM) interferon beta-1a
* Participation in a non-interventional or interventional clinical study of Biogen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RRMS, who are currently stable on a SC interferon beta treatment for at least three months and maximum four years (switch between SC interferon beta treatments possible) will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at Least one Injection Site Reaction (ISR) as Reported by the Participants | Day 1
  ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus.
Percentage of Participants with at Least one Flu-like Symptoms (FLS) as Reported by the Participants | Day 1
  Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.

SECONDARY OUTCOMES:
Percentage of Participants with at Least one ISR (FLS) as Reported by the Nurse | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Percentage of Participants with at Least one ISR (FLS) as Reported by the Physician | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Percentage of Participants with Types of ISR (FLS) Reported by Participants, Nurses, and Physician | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Duration of ISR (FLS) Reported by Participants, Nurses, and Physician | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Usual Time of Occurrence of ISR (FLS) as Reported by the Participants, Nurses and Physicians | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Interference Score of ISR (FLS) With Participant's Daily Activities | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. Interference of ISR (FLS) with participant's daily activities will be assessed by a visual analogue scale ranging from '0' (not at all) to '10' (extremely).
Number of Participants Taking Treatments/Actions to Relieve the ISR (FLS) Assessed by Participants, Nurses and Physicians | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Percentage of Participants With at Least one Self-administered Treatment/Action Resulting in Disappearance or Relief of ISR/FLS | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Percentage of Participants With Reducing or Increasing Frequency of ISR/FLS Compared to Previous Therapy | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.
Percentage of Participants With Reducing or Increasing Intensity of ISR/FLS Compared to Previous Therapy | Day 1
  ISR (FLS) denote events regarding ISR which will be evaluated for FLS simultaneously. ISRs include symptoms like redness, pain, heat, swelling, hematoma (bruising), induration (hardness), blistering, itching, burning, a sore or pus. Flu-like symptoms are specified by fever, chills, aching limbs, headache, sweating, fatigue or weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No